CLINICAL TRIAL: NCT02604121
Title: Interest of Cytological Screening for Early Diagnosis of Precancerous or Cancerous Lesions of Oral Cavity by Transepithelial Brushing in Liquid-based
Brief Title: Cytological Screening for Early Diagnosis of Precancerous or Cancerous Lesions of Oral Cavity
Acronym: Cytobuccale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 12 045 03
Record Dates: First submitted 2015-08-18; First posted 2015-11-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Mouth Neoplasms
Keywords: oral cavity; cancerous and precancerous lesions
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transepithelial brushing (Experimental): transepithelial brushing in liquid-based technology + biopsy
  Interventions: Device: Orcellex® Rovers brush

INTERVENTIONS:
Device: Orcellex® Rovers brush — transepithelial brushing

SUMMARY:
Prospective study of diagnosis validation of a cytological technique. 200 patients with oral cavity cancerous and precancerous lesions will be enrolled.

A cytological sample of the lesion will be performed by transepithelial brushing ( Orcellex® Rovers brush) in cytology liquid-based technology (methode ThinPrep 2000 (Hologic®)). A microscopic double blind reading will be performed. A biopsy sampling will be carried out in accordance with current strategy of screening. The brushing diagnosis quality will be compared to the biopsy which is the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* one or several cancerous or pre-cancerous lesions of oral cavity newly diagnosed or detected during a follow-up visit

Exclusion Criteria:

* pregnant or lactating women
* patients under juridical protection

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic validity of lesion (Bethesda system, 2001) | baseline
  Diagnostic validity (specificity and sensibility, the classification of lesions is performed according Bethesda system, 2001 and the reference is the histology of biopsy of lesion

SECONDARY OUTCOMES:
Diagnostic validity - predictive value (positive and negative) | baseline
  Calculation of predictive value (positive and negative) of cytology / the reference is histology of biopsy
Feasibility of cytology | Baseline
  sample rate not satisfactory= hemorrhage hiding the cells of interest
Feasibility of cytology | Baseline
  sample rate not satisfactory : low cellularity of the material
Reproducibility intra and inter observers (coefficient of kappa de cohen) | Baseline
  reproducibility intra and inter observers of cytology interpretation (kappa de cohen)

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia COLIN-LACOSTE, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France